CLINICAL TRIAL: NCT00796731
Title: A Dose-escalation, Safety and Pharmacokinetic Study of SAR3419 Administered as a Single Agent by Intravenous Infusion Once Weekly in Patients With Relapsed/Refractory CD19-positive B-cell Non-Hodgkin's Lymphoma (NHL)
Brief Title: SAR3419 Administered Weekly in Patients With Relapsed/Refractory CD19-positive B-cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TED6829; EudraCT 2007-004868-41
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Lymphoma; Non-Hodgkin
Keywords: B-cell lymphoma; NHL
MeSH Terms: conditions — Lymphoma; Lymphoma, B-Cell | interventions — coltuximab ravtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: SAR3419 — administered by intravenous infusion

SUMMARY:
The primary objective is to determine the maximum tolerated dose (MTD) of SAR3419 according to the dose limiting toxicities (DLTs) observed when administered as a single agent once weekly.

Secondary objectives are:

* to characterize the global safety profile
* to evaluate the pharmacokinetic (PK) profile of SAR3419 in the proposed dosing schedule
* to assess preliminary evidence of anti-lymphoma activity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of B-cell non Hodgkin's lymphoma
* Relapsed or refractory after standard treatments and with no curative option with conventional therapy (Patients having undergone stem cell transplantation may be included)
* CD19 positive disease by flow cytometry or immunohistochemistry

Exclusion Criteria:

* Burkitt's lymphoma, Lymphoblastic lymphoma, Chronic lymphocytic leukemia (Small lymphocytic lymphoma may be included)
* Evidence of cerebral or meningeal involvement by lymphoma
* Patients without bi-dimensionally measurable disease
* ECOG performance status > 2
* Life expectancy less than 3 months
* Chemotherapy or radiation therapy or other investigational agents within 4 weeks prior to entering the study
* Previous radioimmunotherapy within 12 weeks
* Known anaphylaxis to infused proteins
* HIV, HBV and HCV positivity
* Poor kidney, liver and bone marrow functions
* Any serious active disease or co-morbid condition, which, in the opinion of the principle investigator, will interfere with the safety or the compliance with the study
* Pregnant or breast-feeding women
* Patients with reproductive potential without effective birth control methods

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2008-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Incidence of DLT(s) at each dose level | during the initial 3-week period of treatment

SECONDARY OUTCOMES:
Cumulative DLT(s) | over the entire period of treatment
Incidence of Adverse Events and laboratory abnormalities | study period
Tumor response (complete response, partial response) and duration of the response | study period
Pharmacokinetics parameters | Study period

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand COIFFIER, Professor of Hematology, Principal Investigator — Centre Hospitalier Lyon Sud, France
Locations (6):
- France (6):
  - Sanofi-Aventis Investigational Site Number 250004, Créteil
  - Sanofi-Aventis Investigational Site Number 250006, Lille
  - Sanofi-Aventis Investigational Site Number 250001, Pierre-Bénite
  - Sanofi-Aventis Investigational Site Number 250005, Rennes
  - Sanofi-Aventis Investigational Site Number 250003, Rouen
  - Sanofi-Aventis Investigational Site Number 250002, Villejuif